CLINICAL TRIAL: NCT02887365
Title: A Phase II Study of Tegafur-Uracil as Maintenance Chemotherapy in Patients With Stage II Microsatellite-Stable or Low-Level Microsatellite-Instability Colon Cancer
Brief Title: A Phase II Study of Tegafur-Uracil as Maintenance Chemotherapy in Patients With Stage II of Colon Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 201407054MINC
Record Dates: First submitted 2016-08-01; First posted 2016-09-02 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: MSI-L/MSS; Stage II Colon Cancer
Keywords: colon cancer; MSI-L; MSS; Tegafur-Uracil; Low-Level Microsatellite-Instability
MeSH Terms: conditions — Colonic Neoplasms | interventions — Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tegafur-uracil (Experimental): tegafur-uracil treatment in patients with stage II MSI-L or MSS colon cancer
  Interventions: Drug: tegafur-uracil
- Observation (No Intervention): Observation for one year

INTERVENTIONS:
Drug: tegafur-uracil
  Arms: tegafur-uracil

SUMMARY:
Investigators would like to assess the efficacy and safety of tegafur-uracil in patients with stage II MSI-L or MSS colon cancer under metronomic setting for one year.

DETAILED DESCRIPTION:
Approximately 15% cases of colon cancer are associated a type of inherited susceptibility called defective DNA mismatch repair (MMR), which is frequently measured by either the presence of microsatellite instability (MSI) or by testing for loss of the protein products for genes involved in DNA MMR (MLH1, MSH2, MSH6 and PMS2). Tumors are classified according to the percentage of abnormal microsatellite regions present: >30-40% as high-level MSI (MSI-H), <30-40% as low-level MSI (MSI-L) and no abnormalities as microsatellite stable (MSS). In the condition of MSI presence, evidence shows that MSI is a marker of a more favorable survival outcome and a predictor of decreased benefit from adjuvant therapy with 5-FU in patients with stage II disease. MSI status can be used in the clinic as a prognostic tool to identify a subgroup of stage II patients with improved prognosis. Patients with MSI-H tumors are not suggested to have adjuvant chemotherapy while patients with MSI-L or MSS tumors can benefit from adjuvant chemotherapy. oral tegafur-uracil as an adjuvant chemotherapy in patients with Dukes' stage B2 and C2 colon cancer could be a good alternative to infusional 5-FU. Current evidences suggest adjuvant 5-FU-based therapy could improve survival outcome for patients with stage II MSI-L or MSS colon cancer, but not for patients with MSI-H colon cancer. Thus, oral tegafur-uracil is considered to have similar efficacy as 5-FU in this population.

ELIGIBILITY:
Inclusion Criteria

To be eligible for inclusion, each subject must fulfill all of the following criteria:

1. pathologically confirmed adenocarcinoma of the colon with stage II disease;
2. complete resection of primary tumor;
3. detection of low level microsatellite instability (MSI-L) or microsatellite stable (MSS) in resected tumor sample;
4. no prior chemotherapy or radiotherapy for colon cancer;
5. ECOG performance status 0 to 1;
6. age of 20 years or older;
7. able to start the study treatment within 8 weeks after surgery;
8. able to understand and willingness to sign a written informed consent document.

Exclusion Criteria

Subjects who fulfill any of the following criteria will be excluded from the trial:

1. Severe postoperative complications;
2. inadequate hematopoietic function which is defined as below:

   1. hemoglobin < 9 g/dL;
   2. absolute neutrophil count (ANC) ≤ 1,500/mm3;
   3. platelet count < 100,000/mm3;
3. inadequate hepatic function which is defined as below:

   1. total bilirubin > 2 times upper limit of normal (ULN);
   2. hepatic transaminases (ALT and AST) > 2.5 x ULN;
4. inadequate renal function which is defined as below:

   a.creatinine > 1.5 x ULN;
5. significant medical conditions that is contraindicated to study medication or render patient at high risk from treatment complications based on investigator's discretion;
6. other malignancy within the past 5 years except for adequately treated basal or squamous cell skin cancer or cervical cancer in situ;
7. participation in another clinical trial with any investigational drug within 30 days prior to entry;
8. pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential. Patients with childbearing potential should have effective contraception for both the patient and his or her partner during the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival Safety profile of tegafur-uracil | 3 years
  To observed safety profile of tegafur-uracil as maintenance chemotherapy in patients with stage II microsatellite- stable or low-level microsatellite -instability colon cancer.
  The hematological and biochemistry test should be closely monitored during the treatment period because of bone marrow depression, liver dysfunction, dehydration, anorexia, nausea, vomiting, and other adverse reactions have reported in clinical treatment. The evaluation would be included the date or symptoms that the package insert have mentioned.

SECONDARY OUTCOMES:
5-year overall survival | 3 years
  3-year disease free survival (DFS) rate CT/MRI scan will be performed within 28 days prior to treatment, and then every 4 months from the start of treatment for the 1st year, then every half year for the 2nd year, and every year for the 3rd to 5th year. DFS will be measured from the start date of study treatment to the date of disease recurrence. 5-year overall survival (OS) rate OS will be measured from the start date of study treatment to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Been Ren Lin, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan